CLINICAL TRIAL: NCT05530382
Title: Comparing Self-guided Learning (Video and hands-on Simulation) With Traditional Instructor-led Learning for Medical Device Training: a Randomized-controlled Trial
Brief Title: Self-guided vs Traditional Instructor-led Learning for Medical Device Training
Acronym: EVALUATING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Videolearning
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Professional Role; Interprofessional Education; Simulation Training; Learning Problem
Keywords: Teaching Methods; Learning Methods; Self-Directed Learning; Continuing Medical Education

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- self-guided learning (video and hands-on simulation) (Experimental): video-based self-directed learning
  Interventions: Other: self-guided learning
- traditional instructor-led learning (No Intervention): traditional instructor-led learning in face-to-face workshop

INTERVENTIONS:
Other: self-guided learning — video-based self-directed learning for medical device training
  Arms: self-guided learning (video and hands-on simulation)

SUMMARY:
The aim of this study project is to clarify whether defined practical application skills are learned by anesthesiology specialists through a self-directed learning program with learning videos and a hands-on exercise station ("intervention group"). "Control group" is a traditional instructor-led practical workshop classroom teaching.

Hypothesis: A video-based and self-directed learning program shows no difference in the learning successes than traditional face-to-face workshops.

DETAILED DESCRIPTION:
The Department of Anaesthesiology and Pain Medicine is going to buy and introduce a new generation of anaesthetic machines. Therefore the whole clinical staff of the department who will operate the new anaesthetic machine in the future must be educated and trained with this device before working with patients.

Continuous professional training in the use of medical devices is an essential part of developing professional skills, including in anaesthesia. The professional, routine use of devices is essential to guarantee patient safety. The usual instructor-led workshop-based equipment training in face-to-face lessons is time-consuming and resource-intensive. The high work intensity and shift work in anaesthesia pose a challenge for such training courses. Video-supported learning sequences were more effective than traditional face-to-face lessons, especially for procedural - cognitive processes of complex psychomotor skills. Self-controlled practical practice is more effective than externally controlled practice conditions.

The aim of this study is to clarify whether defined practical application skills (anaesthetic machine) are learned by anesthesiology specialists (nurses and physicians of the department) through a self-directed learning program with learning videos and a hands-on exercise station ("intervention group"). "Control group" is a traditional instructor-led practical workshop classroom teaching.

• The null hypothesis (H0) is that a video-based and self-directed learning program shows no difference in the learning success than traditional face-to-face workshops

The aim of this study is to clarify whether anesthesiologists and nurses anaesthetists can learn defined practical application skills through a self-directed learning program with learning videos and a hands-on training station. If this educational research project is able to demonstrate that self-guided learning of complex psychomotor skills needed for the handling of medical devices like respirators is non-inferior to traditional classroom teaching of such skills, this might minimize the dependence on traditional educator-driven resource-intensive workshop teaching and has the potential to change clinical teaching in the future. The educational topic of the study is "device training in the hospital sector".

A randomized controlled comparative study with two groups (face-to-face workshop versus video-based self-directed learning) in a non-inferiority design is planned, assuming a non-inferior success rate of the traditional face-to-face workshop of 80% and a non-inferiority range of 10%. According to a sample size calculation, 224 voluntary participants are needed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical working anaesthesia staff of the Department of Anaesthesia and Pain Medicine, Bern University Hospital
* written consent

Exclusion Criteria:

- not fulfilling inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Application skills achieved in the context of an objective structured clinical examination (OSCE) test station per participant (yes or no) | 10 minutes
  Achieved or not achieved based on defined practical assignments and oral questioning using a defined catalogue of questions. The testing is carried out by an expert trained as a key user. The test is rated as successful if 60% or more of the questions are answered successfully.
  The following four criteria are checked:
  * Working principle
  * Security aspect
  * Handling and operation
  * Theory-practice transfer
  Each criterion is assessed with 0-3 points 0 = does not apply
  1. = rather does not apply
  2. = applies
  3. = applies very well
  The final evaluation of the device test is based on the following granulated scale:
  A - 100% of the criteria (excellent) B 90% - 99% (very good) C 80% - 89% (good) D 70% - 79% (satisfactory) E 60% - 69% (sufficient) F <60% (unsatisfactory)

SECONDARY OUTCOMES:
level of application skills | 10 minutes
  Application skills scaled (excellent (A) to unsatisfactory (F), measured from the data from the test station.
  The final evaluation of the device test is based on the following granulated scale:
  A - 100% of the criteria (excellent) B 90% - 99% (very good) C 80% - 89% (good) D 70% - 79% (satisfactory) E 60% - 69% (sufficient) F <60% (unsatisfactory)
open questions after the training | 1 day
  Participants will report in a survey if they have any unanswered questions after the training. The number (n) of unanswered questions and percentages will be given for each arm
Time spent | 1 day
  Participants will report in a survey on their time spent for learning. Time will be reported in minutes for each arm per participant.
use of resources | 1 day
  Use of resources in both teaching formats (e.g., books, internet, other teaching material). The outcome will be reported in numbers and percentages.
cost comparison | 1 day
  Cost comparison between the two learning formats. For traditional learning e.g. cost for the instructor and facility. For video-guided learning e.g. costs for the production of the video. The outcome will be reported in Swiss Francs.

CONTACTS AND LOCATIONS:
Overall Officials: Greif Robert, MD, MME, Professor, Study Director — University of Berne; Caterina Gutersohn, RN, NA, Principal Investigator — University of Berne
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Inselspital, Bern University Hospital, University of Bern, Bern, Switzerland, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
All relevant data will be published

REFERENCES:
- [Derived] Gutersohn C, Schweingruber S, Haudenschild M, Huber M, Greif R, Fuchs A. Self-directed learning versus traditional instructor-led learning for education on a new anaesthesia workstation: a noninferiority, randomised, controlled trial. Br J Anaesth. 2025 Oct;135(4):990-996. doi: 10.1016/j.bja.2025.03.043. Epub 2025 May 22. PMID 40410098
- [Derived] Gutersohn C, Schweingruber S, Haudenschild M, Huber M, Greif R, Fuchs A. Medical device education: study protocol for a randomised controlled trial comparing self-directed learning with traditional instructor-led learning on an anaesthesia workstation. BMJ Open. 2023 Sep 4;13(9):e070261. doi: 10.1136/bmjopen-2022-070261. PMID 37666557